CLINICAL TRIAL: NCT04246398
Title: FMT in Children With Autism and Gastrointestinal Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf Harofeh MC (Other Government)
Responsible Party: Sponsor-Investigator, Assaf Harofeh MC, Dr.Ilan Youngster, Head, The Center for Translational Microbiome Research at Shamir Medical Center, Assaf-Harofeh Medical Center
Organization: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0052-19-ASF
Record Dates: First submitted 2020-01-06; First posted 2020-01-29 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Children With Autism
Keywords: Fecal microbiota transplant; autism spectrum disorder; children
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal microbiota transplant (FMT) (Experimental): 10 capsules per dose for 6 consecutive weeks, twice a week, for a total of 120 capsules.
  Each inoculum will be prepared from the feces of 1 donor and a dose of 10 capsules contains sieved, concentrated material derived from a mean of 10 grams of fecal matter. Donors are healthy, nonpregnant adults aged 18 to 50 years, taking no medications, and with a normal body mass index (18.5-25 [calculated as weight in kilograms divided by height in meters squared]).
  Interventions: Other: FMT
- placebo (Placebo Comparator): Placebo capsules will consist of a combination of saline/glycerol (same vehicle as FMT capsules). The inner capsules is dark (green colored), so the general appearance of the capsules is the same to the people who do not prepare them.
  Interventions: Other: FMT - placebo

INTERVENTIONS:
Other: FMT — Participants will be asked to fast for 4 hours prior to and 1 hour following capsule intake.
  Each capsule will be taken with a sip of water, Capsules must not be crushed, chewed, or dissolved Participants will be evaluated for 15 minutes immediately following capsule administration.
  Other Names: Fecal microbiota transplant
  Arms: Fecal microbiota transplant (FMT)
Other: FMT - placebo — Participants will be asked to fast for 4 hours prior to and 1 hour following capsule intake.
  Each capsule will be taken with a sip of water, Capsules must not be crushed, chewed, or dissolved Participants will be evaluated for 15 minutes immediately following capsule administration.
  Arms: placebo

SUMMARY:
1. ASD children with gastrointestinal problems that interfere with daily routine will be recruited at the center for Autism led by Prof Zachor, and at the Pediatric Neurology & Development Center at Shamir Medical Center. Publications in the social media- facebook and support groups for Autism will also be used. The decision whether or not to initiate any medical treatment will not be influenced by the study investigators and will be made solely by the treating doctor.
2. If possible, participants will provide informed consent after receiving a thorough explanation by the study team, as will both parents or other legal guardians.
3. Two groups randomization will be performed, group A and group B. The group randomization will be double blinded.
4. Participants randomized to group A will receive 10 capsules FMT twice a week for 3 weeks, and at week 12 followed by 3 weeks placebo twice a week.
5. Participants randomized to group B will receive 10 capsules placebo twice a week for 3 weeks and at week 12 followed by 3 weeks FMT twice a week.
6. At baseline, participants will undergo a full physical examination, vital signs, medical questionnaire, ROME III questionnaire for kids >age4 />age 10, ATN-GISSI-17 questionnaire, Aut-Eat questionnaire regarding eating habbits, the Social Responsiveness Scale (SRS) and the Adaptive Behavior Assessment System (ABAS).
7. Parents/ care providers will fill a daily symptoms follow-up questionnaire at baseline
8. Fecal samples will be provided for analysis of microbiome and proteome at beseline, weeks 3,12, 15 and 6+9 months.
9. At each FMT/Placebo administration a short questionnaire asking about possible adverse events, GI symptoms, overall well-being, and medication changes will be administered

DETAILED DESCRIPTION:
About 50% of children with Autism spectrum disorder (ASD) tend to suffer from one or more gastrointestinal (GI) symptoms.The GI symptoms vary from constipation (~20%), diarrhea (~14%), Abdominal pain/discomfort (14%), bloating (12%), incontinence (12%), reflux (7.4%), nausia (6%) and difficult with bowel movements (6%).

The severity of ASD is associated with the observed GI symptoms, although no cause-effect relationship between GI symptoms and ASD was proven so far. ASD with GI symptoms patients might display significant behavioral manifestations, such as anxiety, self-injury and aggression and these may be attributed to the GI symptoms themselves. Therefore alleviation of the GI symptoms could be important also for improvement of ASD.

In addition to the possibility that the nervous system influences the gut and the GI symptoms, there is also the possibility that the gut and the microbiome within the gut may influence the central nervous system.

Considering the findings that children with ASD have a history of using significantly more antibiotics and that gut permeability increases in ASD it is reasonable to assume that ASD patients have distinct microbiomes and gut metabolites.

Nevertheless, perhaps changing the gut microbiome could lead to improvement in some of the symptoms. So far, studies on influencing ASD (behavior and GI symptoms) by addressing the gut microbiome are optimistic but mostly open-labeled and still inconclusive.

ELIGIBILITY:
Inclusion Criteria:

* ASD Boys or girls 7 - 20 years of age
* suffering gastro-intestinal symptoms and/or food selectivity that interfere with daily routine
* Patients not started on immune-suppressive or anti-inflammatory medications.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women of childbearing potential will have a urine pregnancy test, which must be negative, on Study Day 1, prior to receiving FMT. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for 3 months after FMT.
* Hasn't taken antibiotics 2 days prior to 1st visit.
* Ability of parents or other legal guardian to understand and the willingness to sign a written informed consent document, including the willingness to accept risk of unrelated donor stool.
* Ability to swallow oral medications.

Exclusion Criteria:

* Severe GI problems that require immediate treatment (life-threatening).

  * recent/scheduled surgeries
  * diagnosed as severely malnourished or underweight
  * diagnosed with a single-gene disorder
  * major brain malformations
  * inflammatory bowel diseases
  * known positive serology for celiac disease or eosinophilic esophagitis
  * Pregnancy / breast-feeding
  * Using immune-suppressive or anti-inflammatory medications
  * Active or uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
  * Delayed gastric emptying syndrome
  * Known chronic aspiration
  * History of significant allergy to foods
  * Unable to swallow pills

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 3 weeks from the start of the study
  The safety of using FMT capsules in autistic children with gastrointestinal symptoms is measured by the prevalence and severity of side effects that occurred after taking the capsules, and were documented in a daily follow-up questionnaire
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | 15 weeks from the start of the study
  The safety of using FMT capsules in autistic children with gastrointestinal symptoms is measured by the prevalence and severity of side effects that occurred after taking the capsules, and were documented in a daily follow-up questionnaire
Significant change in GI symptoms [efficiency] | 3 weeks from the start of the study
  effectiveness of FMT capsules in alleviation of GI symptoms in Autistic children is defined by a significant change in the Rome III questionnaire, used for diagnostic of pediatric functional GI disorders
Significant change in GI symptoms [efficiency] | 15 weeks from the start of the study
  effectiveness of FMT capsules in alleviation of GI symptoms in Autistic children is defined by a significant change in the Rome III questionnaire, used for diagnostic of pediatric functional GI disorders
Significant change in GI symptoms [efficiency] | 6 months from the start of the study
  effectiveness of FMT capsules in alleviation of GI symptoms in Autistic children is defined by a significant change in the Rome III questionnaire, used for diagnostic of pediatric functional GI disorders
Significant change in GI symptoms [efficiency] | 9 months from the start of the study
  effectiveness of FMT capsules in alleviation of GI symptoms in Autistic children is defined by a significant change in the Rome III questionnaire, used for diagnostic of pediatric functional GI disorders

SECONDARY OUTCOMES:
Change in food selection [efficiency] | 12 weeks from the start of the study
  The effectiveness of FMT capsules on food selectivity in autistic children is measured using a eating habits questionnaire (Aut-Eat)
Change in food selection [efficiency] | 6 months from the start of the study
  The effectiveness of FMT capsules on food selectivity in autistic children is measured using a eating habits questionnaire (Aut-Eat)
Change in food selection [efficiency] | 9 months from the start of the study
  The effectiveness of FMT capsules on food selectivity in autistic children is measured using a eating habits questionnaire (Aut-Eat)
Improving ASD symptoms [efficiency] | 3 months from the start of the study
  The efficacy of FMT capsules in improving ASD symptoms is measured using the SRS questionnaire (Social Responsiveness Scale) The Total Score calculated separately for males and females. It can be expressed as a raw score or a T-score.
Improving ASD symptoms [efficiency] | 6 months from the start of the study
  The efficacy of FMT capsules in improving ASD symptoms is measured using the SRS questionnaire (Social Responsiveness Scale) The Total Score calculated separately for males and females. It can be expressed as a raw score or a T-score.
Diversity and variability of the gut microbiome | 3 weeks from the start of the study
  Changing the diversity and variability of the gut microbiome measured by sequencing the 16's rRNA.
Diversity and variability of the gut microbiome | 12 weeks from the start of the study
  Changing the diversity and variability of the gut microbiome measured by sequencing the 16's rRNA.
Diversity and variability of the gut microbiome | 15 weeks from the start of the study
  Changing the diversity and variability of the gut microbiome measured by sequencing the 16's rRNA.
Diversity and variability of the gut microbiome | 3 months from the start of the study
  Changing the diversity and variability of the gut microbiome measured by sequencing the 16's rRNA.
Diversity and variability of the gut microbiome | 6 months from the start of the study
  Changing the diversity and variability of the gut microbiome measured by sequencing the 16's rRNA.

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf-HarofehMC, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No